CLINICAL TRIAL: NCT03870789
Title: Field Paramedic Application of Sepsis Triage
Acronym: FAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 3075-C
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Sepsis
Keywords: sepsis, septic shock, early warning scores, infecion
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: The Investigators will examine data from 1-year prior to paramedic implementation of the Hamilton Early Warning Score tool.
- Prospective: The Investigators will examine data from 1-year after paramedic implementation of the Hamilton Early Warning Score tool.

SUMMARY:
Given the implementation of the Hamilton Early Warning Score (HEWS) and the use of capnography by paramedics, this study will involve a large multi-site retrospective evaluation (before vs after implementation) of the HEWS score and comparison of the HEWS to systemic inflammatory response syndrome (SIRS), quick Sepsis Related Organ failure Assessment (qSOFA) and Modified Early Warning Score (MEWS) when applied retrospectively for the identification of sepsis in the prehospital setting.

DETAILED DESCRIPTION:
1. To determine the accuracy of the HEWS score, compared to qSOFA, and SIRS for early sepsis recognition when used in the prehospital setting by paramedics for the identification of patients with sepsis or suspected sepsis.
2. To evaluate the addition of ETCO2 values to predict mortality in patients who screen positive for sepsis.
3. To identify the before and after healthcare outcomes of a prehospital sepsis alert program.

ELIGIBILITY:
Inclusion Criteria:

Any patient to which paramedics apply the Hamilton Early Warning Score or patients who arrive to the Emergency Department (ED) by ambulance without a pre-alert and meet the definition of sepsis in the ED will also be included, and patient is ≥ 18 years

Exclusion Criteria:

Patient is an inter-facility transfer, or patients with absent vital signs are absent, or death before blood can be drawn in the Emergency Department, or the patient fits the criteria for another prehospital alert (ST-elevation myocardial infarction, cerebrovascular vascular accident, or trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-12-11 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of HEWS | 1 year
  To determine the accuracy of the HEWS score, compared to qSOFA, and SIRS for early sepsis recognition when used in the prehospital setting by paramedics for the identification of patients with sepsis or suspected sepsis.

SECONDARY OUTCOMES:
Evaluate the addtion of end-tidal carbon dioxide (ETCO2) values | 1 year
  To evaluate the addition of ETCO2 values to predict mortality in patients who screen positive for sepsis.
Evaluate sepsis alert program | 2 years
  To identify the before and after healthcare outcomes of a prehospital sepsis alert program.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Wellsford, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Centre for Paramedic Education and Research, Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Canadian Institute for Health Information. In Focus: A National Look at Sepsis.; 2009. https://secure.cihi.ca/free_products/HSMR_Sepsis2009_e.pdf.
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675